CLINICAL TRIAL: NCT00085371
Title: A Phase II Study Of Triapine For Advanced Adenocarcinoma Of The Pancreas
Brief Title: Triapine as First-Line or Second-Line Therapy in Treating Patients With Locally Advanced or Metastatic Cancer of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01452; NCI-2012-01452 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-MC0345; CDR0000368762; NCI-6293; MC0345 (Other: Mayo Clinic); 6293 (Other: CTEP); N01CM62205 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

ARMS (1):
- Treatment (triapene) (Experimental): Patients receive triapene IV over 2 hours on days 1-4 and 15-18. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: triapine

INTERVENTIONS:
Drug: triapine — Given IV

SUMMARY:
This phase II trial is studying how well triapine works as first-line or second-line therapy in treating patients with locally advanced or metastatic adenocarcinoma (cancer) of the pancreas. Drugs used in chemotherapy, such as triapine, work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the 3- and 6-month survival rate of patients with locally advanced or metastatic adenocarcinoma of the pancreas treated with 3-AP (Triapine^®) as first- or second-line therapy.

SECONDARY OBJECTIVES:

I. Determine the toxicity and tolerability of this drug in these patients. II. Determine the time to treatment failure in patients treated with this drug. III. Determine overall survival and disease progression in patients treated with this drug.

IV. Determine tumor response in patients treated with this drug. V. Determine laboratory studies that will increase our understanding of Triapine and its effects on cellular processes.

OUTLINE: This is a multicenter study. Patients are stratified according to prior chemotherapy (yes vs no).

Patients receive triapene IV over 2 hours on days 1-4 and 15-18. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3-6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Unresectable disease
  * Locally advanced or metastatic disease
* At least 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan

  * Measurable lesions outside prior radiotherapy field OR measurable lesions actively growing in the site of prior radiotherapy
* No prior chemotherapy OR previously treated with 1, and only 1, gemcitabine-containing regimen for metastatic, unresectable, or locally advanced pancreatic cancer

  * Adjuvant therapy not considered prior chemotherapy if all treatment was completed > 6 months before tumor recurrence
* No known brain metastases
* Performance status - ECOG 0-2
* At least 6 weeks
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 75,000/mm^3
* AST =< 3 times upper limit of normal (ULN)
* Bilirubin =< 1.5 times ULN
* Creatinine =< 1.5 times ULN
* Creatinine clearance > 60 mL/min
* No uncontrolled congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No pulmonary disease requiring oxygen
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No glucose-6-phosphate dehydrogenase (G6PD) deficiency (for patients of African, Asian, or Mediterranean origin or ancestry)
* No active or ongoing infection
* No hypersensitivity or severe allergic reaction to 3-AP (Triapine®) or related compounds
* No concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent antineoplastic therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational therapy for the malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2004-07; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Survival in patients receiving triapine as first-line therapy | 6 months
  The point estimate of the success rates will be calculated as the number of successes divided by the number of evaluable patients, with confidence intervals calculated by the method of Duffy and Santner.
Survival in patients receiving triapine as second-line therapy | 4 months
  The point estimate of the success rates will be calculated as the number of successes divided by the number of evaluable patients, with confidence intervals calculated by the method of Duffy and Santner.

SECONDARY OUTCOMES:
Incidence of adverse events assessed using CTCAE version 3.0 | Up to 3 years
Time to treatment failure | Time from the date of randomization to the date at which the patient is removed from treatment due to progression, toxicity, or refusal, assessed up to 3 years
Overall survival | Up to 3 years
Time to disease progression | Time from registration to documentation of disease progression, assessed up to 3 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Confirmed tumor response, defined to be a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart | 6 months (first 6 courses of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Holen, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States